CLINICAL TRIAL: NCT02196207
Title: Phase III INHIBIT Platform: Prevention Trial, Eloctate vs Emicizumab to Prevent Inhibitors; Eradication Trial: Eloctate Immune Tolerance (ITI) Plus Emicizumab vs vs Eloctate ITI Alone to Eradicate Inhibitors in Severe Hemophilia A
Brief Title: Hemophilia Inhibitor Clinical Trials (INHIBIT) Platform
Acronym: INHIBIT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was revised to be two protocols, one Prevention, one Eradication Trials.
Sponsor: Margaret Ragni (Other)
Responsible Party: Sponsor-Investigator, Margaret Ragni, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO14020038
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Severe Hemophilia A
Keywords: Severe Hemophilia A; Hemophilia Inhibitor Formation; Eloctate; Emicizumab; Inhibitor Prevention; Inhibitor Eradication
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Intervention Model Description: Two phase III randomized trials, each with two arms, including one inhibitor prevention trial and one inhibitor eradication trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Eloctate Prophylaxis (Experimental): Prevention Trial, Arm A: rFVIIIFc (Eloctate) 65 IU/kg weekly will be administered by intravenous infusion in previously untreated children with severe hemophilia A beginning before the first bleed and continued for up to 48 weeks.
  Interventions: Drug: Eloctate Prophylaxis
- Emicizumab Prophylaxis (Experimental): Prevention Trial, Arm B: Emicizumab 1.5 mg/kg weekly (following 4-wk induction at 3 mg/kg weekly) will be administered by subcutaneous injection in previously untreated children with severe hemophilia A beginning before the first bleed and continued for up to 48 weeks.
  Interventions: Drug: Emicizumab Prophylaxis
- Eloctate ITI plus Emicizumab (Experimental): Eradication Trial, Arm A: Eloctate 100 IU/kg every other day will be administered by intravenous infusion as immune tolerance plus Emicizumab 1.5 mg/kg weekly by subcutaneous injection in previously treated children and adults with severe hemophilia A and high-titer inhibitors and continued for up to 48 weeks.
  Interventions: Drug: Eloctate ITI plus Emicizumab
- Eloctate ITI Alone (Active Comparator): Eradication Trial, Arm B: Eloctate 100 IU/kg every other day will be administered by intravenous infusion as immune tolerance alone in previously treated children and adults with severe hemophilia A and high-titer inhibitors and continued for up to 48 weeks.
  Interventions: Drug: Eloctate ITI

INTERVENTIONS:
Drug: Eloctate Prophylaxis — Prevention Trial, Arm A: Eloctate (65 IU/kg) will be administered weekly by intravenous infusion for up to 48 weeks in previously untreated children with severe hemophilia A beginning before the first bleed.
  Other Names: rFVIIIFc Prophylaxis
  Arms: Eloctate Prophylaxis
Drug: Emicizumab Prophylaxis — Prevention Trial, Arm B: Emicizumab (1.5 mg/kg) will be administered weekly by subcutaneous injection for up to 48 weeks in previously untreated children with severe hemophilia A.
  Other Names: Hemlibra Prophylaxis
  Arms: Emicizumab Prophylaxis
Drug: Eloctate ITI plus Emicizumab — Eradication Trial, Arm A: Eloctate (100 IU/kg) ITI every other day by intravenous infusion plus Emicizumab (1.5 mg/kg) weekly by subcutaneous injection will be administered for up to 48 weeks as immune tolerance in children and adults with severe hemophilia A and high-titer inhibitors.
  Other Names: rFVIIIFc ITI plus Hemlibra
  Arms: Eloctate ITI plus Emicizumab
Drug: Eloctate ITI — Eradication Trial, Arm A: Eloctate (100 IU/kg) ITI every other day by intravenous infusion will be administered for up to 48 weeks as immune tolerance in children and adults with severe hemophilia A and high-titer inhibitors.
  Other Names: rFVIIIFc ITI
  Arms: Eloctate ITI Alone

SUMMARY:
This study will evaluate if Eloctate is superior to Emicizumab in reducing inhibitors in children with severe hemophilia when given before the first bleed (preemptive) and continued weekly to prevent bleeds (prophylaxis); and whether Eloctate immune tolerance induction (ITI) plus emicizumab is superior to Eloctate ITI alone in eradicating inhibitor formation in children and adults with severe hemophilia A.

DETAILED DESCRIPTION:
This is a multi-center, randomized Phase III Clinical Trials Platform (INHIBIT) in which hemostatic agents will be compared using adaptive design to prevent and eradicate inhibitors in patients with severe hemophilia A. This adaptive design is necessary as randomized trials in rare diseases are otherwise not possible. The INHIBIT Trial Platform includes one Inhibitor Prevention Trial and one Inhibitor Eradication Trial that will be conducted at up to 41 U.S. hemophilia treatment centers (HTCs) affiliated with universities. The Inhibitor Prevention Trial is a 48-week randomized phase III trial in which 66 previously untreated patients (PUPs) (children < 6 yr) with severe hemophilia A will be enrolled and randomized to preemptive weekly Eloctate vs. Emicizumab to prevent inhibitor formation, defined as anti-FVIII > 5.0 BU. The Inhibitor Eradication Trial is a 48-week randomized phase III trial in which 90 previously-treated patients (PTPs) with severe hemophilia A and high-responding inhibitors (anti-VIII >5.0 B.U.), including subjects developing inhibitors during the Prevention Trials and adults or children of any age at the same HTCs refractory to or never previously tolerated, will be enrolled and randomized to Eloctate ITI god plus weekly Emicizumab vs. Eloctate ITI alone to eradicate inhibitor formation, defined as anti-FVIII<0.6 B.U. Blood draws will be minimized to 6 timepoints, pre, 4, 12, 24, 36, and 48 weeks, and validated for small volumes, 3.8 cc (¾ tsp) each. The Inhibit Trials Platform is considered greater than minimal risk as study drug is given before the first bleed and special inhibitor studies are obtained.

ELIGIBILITY:
Prevention Trial, Inclusion Criteria:

* Male children >/= 4 months of age.
* Severe hemophilia A (FVIII < 0.01 U/ml)
* No previous bleed or surgery requiring treatment (except circumcision)
* No previous factor VIII product (except for circumcision)
* Willingness to comply with weekly prophylaxis for 48 weeks
* Willingness of parent/caregiver to keep a personal diary of bleeding frequency and factor treatment.
* Willingness to make monthly visits and coagulation testing at weeks 4, 12, 24, 36, and 48 (end of study)

Prevention Trial, Exclusion Criteria:

* Acquired hemophilia.
* Any bleeding disorder other than hemophilia A.
* Treatment with clotting factor previously, other than circumcision.
* Presence of an inhibitor to factor VIII.
* Use of an experimental drug(s).
* Surgery anticipated in the next 48 weeks.
* Life expectancy less than 5 years.
* Inability to comply with study requirements.

Eradication Trial, Inclusion Criteria:

* Male adults or children with no age limitation.
* Severe hemophilia A (FVIII <0.01 U/ml).
* Presence of an inhibitor to FVIII (anti-FVIII > 5.0 B.U.)
* Willingness to comply with study drugs for up to 48 weeks.
* Willingness to keep a personal diary of bleed frequency and drug treatment.
* Willingness to make monthly visits and coagulation testing at weeks 4, 12, 24, 36, and 48 (end of study).

Eradication Trial, Exclusion Criteria:

* Acquired hemophilia.
* Any bleeding disorder other than hemophilia A.
* Current use of Emicizumab, or if used, > 8 weeks since last treatment.
* Use of an experimental drug(s).
* Surgery anticipated in the next 48 weeks.
* Life expectancy less than 5 years.
* Inability to copy with study requirements.

Ages: 4 Months to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Prevention Trial: Time to inhibitor formation | Up to 48 weeks
  Inhibitor formation is defined as anti-FVIII > / = 5.0 B.U. by chromogenic Nijmegen-modified Bethesda assay, performed on plasma, repeated for confirmation.
Eradication Trial: Time to inhibitor eradication | Up to 48 weeks
  Inhibitor eradication is defined as anti-FVIII < 0.6 B.U. by chromogenic Nijmegen Bethesda assay, performed on plasma, repeated for confirmation.

SECONDARY OUTCOMES:
Prevention & Eradication Trials: Bleeding events including hematoma, joint, central nervous system, other | Up to 48 weeks
  Number of bleeding events
Prevention & Eradication Trials: Factor VIII trough activity by chromogenic assay | Up to 48 weeks
  FVIII activity
Prevention & Eradication Trials: HLA type and factor VIII genotype | Up to 48 weeks
  HLA haplotype and FVIII mutation

OTHER OUTCOMES:
Prevention & Eradication Trials: T Cell Elispot Assay | Up to 48 weeks
  T cell reactivity to FVIII

CONTACTS AND LOCATIONS:
Overall Officials: Margaret V Ragni, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A biologic specimen and data repository for this trial will be available, pending NHLBI approval, at BioLINCC https://biolincc.nhlbi.nih.gov, to any research or investigator who makes formal application request and is formally approved by NHLBI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year of trial completion.
Access Criteria: Access will be determined by NHLBI.

REFERENCES:
- [Derived] Ragni MV. The effect of emicizumab regimen on haemophilia outcomes. Lancet Haematol. 2019 Jun;6(6):e286-e287. doi: 10.1016/S2352-3026(19)30070-5. Epub 2019 Apr 16. No abstract available. PMID 31003964